CLINICAL TRIAL: NCT02290561
Title: SmartTarget - A Magnetic Resonance Image to Ultrasound Fusion System for Targeted Prostate Intervention: Therapy
Brief Title: SmartTarget THERAPY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/0389
Record Dates: First submitted 2014-11-10; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; Therapeutics; Magnetic Resonance Imaging; Ultrasonography; High Intensity Focused Ultrasound; Image Fusion
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: SmartTarget Therapy — MRI to Ultrasound fusion directed HIFU
Device: MRI
Device: high intensity focused ultrasound (HIFU)

SUMMARY:
The purpose of this study is to assess how accurately SmartTarget can direct high intensity focused ultrasound (HIFU) to a pre-defined area (cancer) in the prostate.

The current standard methods for treating prostate cancer are directed to the whole gland - either surgery to remove it or radiotherapy. An alternative method is focal therapy. This is surgery that uses an energy source to ablate the cancer whilst preserving the normal healthy tissue.

Prior to surgery prostate cancer can often be localised using MRI imaging and detailed prostate biopsy techniques. The difficulty is that during surgery it is very difficult to accurately locate the cancer on the live ultrasound images - to compensate surgeons will treat half or a quarter of the prostate to ensure that the cancer is treated. This may cause higher rates of side-effects.

SmartTarget is an MRI to ultrasound fusion device that maps the pre-treatment MRI onto the live ultrasound during surgery. It then provides a target for the surgeons to treat during the operation.

The results will measure if the area intended to treat was covered and if how accurate the treatment was by comparing the pre-treatment MRI with a 1 week post treatment scan

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of prostate cancer (PSA </=15ng/ml, Gleason score </=4+3, and radiological stage </=T3aNoMo)
2. Prostate biopsy concordant with mpMRI lesion (template transperineal or MRI-targeted biopsy only)
3. Discrete lesion on mpMRI scoring 3, 4 or 5 on radiological scale of suspicion
4. mpMRI carried out according to European Society of Uro-Radiology guidelines at 1.5T or 3T
5. An understanding of the English language sufficient to understand written and verbal information about the trial and consent process
6. Signed informed consent

Exclusion Criteria:

1. No lesion on mpMRI
2. Bilateral lesions on mpMRI
3. mpMRI undertaken over 6 months prior to visit 1
4. Contralateral Gleason >/=3+4 and/or Maximum Cancer Core Length Involvement >/=6mm
5. Men who have taken any form of hormones (except 5-alpha reductase inhibitors) within the last 6 months
6. Prior immunosuppression or predefined immunosuppressed state
7. An irreversible coagulopathy predisposing to bleeding
8. Unable to undergo transrectal ultrasonography
9. Previous radiation therapy to the pelvis
10. Previous HIFU, cryosurgery, thermal, irreversible electroporation, radiofrequency or microwave therapy to the prostate.
11. Men with evidence of metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging
12. Men not fit for major surgery as assessed by a consultant anaesthetist
13. Men who are unable to give informed consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Target Ablation | 1 week post treatment
  The ability of SmartTarget-directed focal HIFU therapy to ablate an intended target within the prostate, as measured by the proportion of men in whom complete ablation of the target region is achieved. Complete or incomplete ablation is determined by a comparative assessment of the pre-therapy and one week post-therapy contrast-enhanced MRIs by an expert radiologist.

SECONDARY OUTCOMES:
Accuracy | 1 week post treatment
  The accuracy of SmartTarget guided focal HIFU measured by the relative treatment volume and relative ablation volume on the one week post treatment.
Length of the procedure | intraoperative
  The efficiency and clinical usability of the SmartTarget device as measured by the:
  Length of the procedure
  The time taken during the procedure using SmartTarget, including:
  The total prostate computer model generation time The total time taken to register (fuse) MRI and ultrasound image data and the number of times an image registration is performed using SmartTarget (the re-registration rate) SmartTarget failure rate
Quality of Life | 6 weeks and 3 months
  To assess how this treqatment strategy impacts on quality of life as measured using validated questionnaires at 6 weeks and 3 months post treatment.
  IPSS IIEF EQ5D - 5L

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, FRCS PhD, Principal Investigator — University College, London